CLINICAL TRIAL: NCT04002674
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Impact of Nilotinib Treatment on Safety, Tolerability, Pharmacokinetics and Biomarkers in Dementia With Lewy Bodies (DLB)
Brief Title: Impact of Nilotinib on Safety, Tolerability, Pharmacokinetics and Biomarkers in Dementia With Lewy Bodies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Fernando Pagan MD, Associate Professor, Department of Neurology Co-Director, Movement Disorders Program Director, NPF Center of Excellence Associate Professor, SOM Clinical Track, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000122
Record Dates: First submitted 2019-04-08; First posted 2019-06-28 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease | interventions — nilotinib

STUDY DESIGN:
Intervention Model Description: Investigators will evaluate the effects of 200 mg of Nilotinib versus matching Placebo taken daily by mouth for 6 Months, followed by 1 Month wash-out period in individuals with DLB.
  Sixty (60) participants will be recruited and randomly assigned 1:1 to placebo (arm 1) or 200 mg Nilotinib (arm 2). Participants will be treated for 6 months and monitored every month (4 weeks) in a total of 9 visits that include screening, baseline, 1, 2, 3, 4, 5, 6 months follow up and 7-month washout.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized by a Biostatistician by an internet based randomization module into two groups. The researchers include : Primary investigator , Sub-Investigators ,Clinical Coordinators, Nurse Practitioners , and Clinical Reseach unit staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Sixty (60) participants will be recruited and randomized into 2 arms (1:1). Thirty (30) patients in arm 1 will receive the matching placebo ("sugar pill") one (1) capsule orally (without food) once daily for 6 months (180 days).
  Interventions: Drug: Placebo oral capsule
- 200 mg Nilotinib (Active Comparator): Sixty (60) participants will be recruited and randomized into 2 arms (1:1). Thirty (30) patients in arm 2 will receive the 200 mg of Nilotinib one (1) capsule orally (without food) once daily for 6 months (180 days).
  Interventions: Drug: Nilotinib Oral Capsule

INTERVENTIONS:
Drug: Placebo oral capsule — Thirty (30) patients in arm 1 will receive the matching placebo ("sugar pill") one (1) capsule orally (without food) once daily for 6 months (180 days).
  Other Names: Placebo
  Arms: Placebo
Drug: Nilotinib Oral Capsule — Thirty (30) patients in arm 2 will receive the 200 mg of Nilotinib one (1) capsule orally (without food) once daily for 6 months (180 days).
  Other Names: Tasigna
  Arms: 200 mg Nilotinib

SUMMARY:
Dementia with Lewy Bodies (DLB) is an alphasynucleinopathy and the second most common form of dementia in the elderly. DLB shares striking neuropathological and clinical similarities with both Parkinson's disease (PD) and Alzheimer's disease (AD). Nilotinib (Tasigna®, AMN107, Novartis, Switzerland) is approved by the FDA and is well tolerated for CML treatment at oral doses of 600-800mg daily. The Investigators propose to perform a phase II randomized, double blinded, placebo controlled study to evaluate the impact of Nilotinib in patients with DLB.

DETAILED DESCRIPTION:
A phase II randomized, double blinded, placebo controlled study will be performed to evaluate the impact of Nilotinib (Tasigna®, AMN107, Novartis, Switzerland) on safety, tolerability, pharmacokinetics, pharmacodynamics and clinical outcomes in patients with Dementia with Lewy Bodies. Sixty ( 60) participants will be recruited and randomly assigned 1:1 to placebo (arm 1) or 200 mg Nilotinib (arm 2).This study will be conducted in DLB patients with 2.5≥Hoehn & Yahr≤3 and UPDRS I-III ≤50 and 15≥UPDRS III (motor) ≥40 (Unified Parkinson's Disease Rating Score)and MoCA≥18(Montreal Cognitive Assessment). Eligible participants must be stable on MAO-B inhibitors (Rasageline or Selegeline) for 4 weeks and must not be on ≥800mg Levodopa daily. Participants must be stable on acetylcholinesterase inhibitors and other medications for at least 6 weeks. Participants will be treated for 6 months and monitored every month ( 4 weeks) in a total of 9 visits that include screening , baseline, 1, 2, 3, 4, 5, 6 months follow up and 7 month washout. Blood and cerebrospinal fluid (CSF) will be collected at baseline and at 6 months to determine Nilotinib effects on CSF biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Capable of providing informed consent and complying with study procedures. Subjects who are unable to provide consent may use a Legally Authorized Representative (LAR).
3. Clinical diagnosis of DLB according to McKeith et al (7) with both dementia MoCA≥18 and Parkinsonian defined as bradykinesia in combination with rest tremor, rigidity or both UPDRS I-III is less than 50 and/or UPDRS-III between 15 -40 on-state. Dementia and Parkinsonism must be present with at least one other symptom such as fluctuation, visual hallucinations or REM sleep behavioral disorder (RBD)
4. 2.5 ≥Hoehn and Yahr stage ≤3
5. MDS-UPDRS-III 15-40 on-state (or up to 70 on the off state)
6. Abnormal DaTScan
7. Stable concomitant medical and/or psychiatric illnesses in the judgement of the PI
8. Patients between the age of 25-90 years, medically stable
9. Must NOT be stable on mono-amine oxidase (MAO)-B inhibitors (Selegeline or rasagiline) for at least 4 weeks before enrollment and during Nilotinib treatment.
10. Must be medically stable on less than or equal to 800mg Levodopa daily for at least 4 weeks
11. QTc interval 350-460 ms, inclusive
12. Participants must be willing to undergo LP at baseline and 6 months after treatment

Exclusion Criteria:

1. Patients with hypokalemia, hypomagnesaemia, or long QT syndrome- QTc≥461 ms
2. Concomitant drugs known to prolong the QTc interval and history of any cardiovascular disease, including myocardial infraction or cardiac failure, angina, arrhythmia
3. History or presence of cardiac conditions including:

   1. Cardiovascular or cerebrovascular event (e.g. myocardial infarction, unstable angina, or stroke)
   2. Congestive heart failure
   3. First, second- or third-degree atrioventricular block, sick sinus syndrome, or other serious cardiac rhythm disturbances
   4. Any history of Torsade de Pointes
4. Treatment with any of the following drugs at the time of screening or the preceding 30 days, and/or planned use over the course of the trial:

   1. Treatment with Class IA or III antiarrhythmic drugs (e.g. quinidine)
   2. Treatment with QT prolonging drugs (www.crediblemeds.org)- excluding Selective Serotonin Reuptake Inhibitors (SSRIs) (e.g. Citalopram, Paxil, Zoloft, Cymbalta, Sertraline, etc...)
   3. Strong CYP3A4 inhibitors (including grapefruit juice). The concomitant use of strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole) must be avoided. Grapefruit products may also increase serum concentrations of Nilotinib. Should treatment with any of these agents be required, therapy with Nilotinib should be interrupted.
   4. Anticoagulants, including Coumadin (warfarin), heparin, enoxaparin, daltiparin, xarelto, etc.
   5. St. John's Wort and the concomitant use of strong other CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital) must be avoided since these agents may reduce the concentration of Nilotinib.
5. Abnormal liver function defined as AST and/or ALT > 100% the upper limit of the normal
6. Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal
7. History of HIV, clinically significant chronic hepatitis, or other active infection
8. Females must not be lactating, pregnant or with possible pregnancy
9. Medical history of liver or pancreatic disease
10. Clinical signs indicating syndromes other than DLB, including, PD, PD with Dementia (PDD), corticobasal degeneration, supranuclear gaze palsy, multiple system atrophy, chronic traumatic encephalopathy, signs of frontal dementia, history of stroke, head injury or encephalitis, cerebellar signs, early severe autonomic involvement, Babinski sign
11. Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
12. Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal or other systemic disease or laboratory abnormality
13. Active neoplastic disease, history of cancer five years prior to screening, including breast cancer (history of skin melanoma or stable prostate cancer are not exclusionary)
14. Contraindications to LP: prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelets < 100,000, use of Coumadin/warfarin, or history of a bleeding disorder
15. Must not be on any immunosuppressant medications or IVIG
16. Must not be enrolled as an active participant in another clinical study

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: occurrence of adverse events (AEs) | 6 Months
  The Investigators will determine safety and tolerability using the occurrence of adverse events (AEs) of interest as per Nilotinib Investigator Brochure (IB).

SECONDARY OUTCOMES:
The Investigator will determine Nilotinib levels in CSF and plasma. | 6 Months
  Pharmacokinetics: Measure the CSF concentration of Nilotinib
The Investigators will determine changes in DLB related CSF and plasma biomarkers | 6 Months
  Pharmacodynamics: Determine the effects of Nilotinib on primary biomarkers, including changes of CSF levels of HVA between baseline and 6 months.Furthermore, measure the CSF concentration of surrogate/exploratory biomarkers.
The investigators will quantify amyloid burden via Florbetaben PET scan | 6 Months
  Quantification of brain amyloid burden via Florbetaben PET at baseline and 6 months (end of treatment)

OTHER OUTCOMES:
Measurement of the effects of Nilotinib on Cognition using the Montreal Cognitive Assessment (MoCA) | 6 Months
  The MoCA is designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains, including attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations and orientation. Scores range between 0 and 30 where 30 is the highest score and 0 is the lowest score.
Measurement of the effects of Nilotinib on Cognition using the Trail Making Test (TMT) | 6 Months
  The Trail Making Test (TMT) is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. The time to complete the test is measured in seconds.
Measuring the effects of NIlotinib on Cognition using the Alzheimer's Disease Assessment Scale - cognitive (ADAS-cog). | 6 Months
  ADAS-cog aims to evaluate cognitive impairment in Alzheimer's disease. ADAS-cog was included in this LBD study to better capture potential changes in activities of daily living (ADL) and non-ADLs and severity of cognitive impairment. Points for errors in each task are added up and the greater the dysfunction, the greater the total score. The lower the dysfunction the lower the total score .
Measuring the effects of Nilotinib on Behavior using the Alzheimer's disease Cooperative Study-Activity of Daily Living scale | 6 Months
  ADCS-ADL is an activity of daily living inventory to assess functional performance. Using a structured interview format, study partners are queried as to whether participants attempted each item in the inventory during the prior 4 weeks and their level of performance. The ADCS-ADL includes some items from traditional basic ADL tests as well as instrumental (complex) activities of daily living. It is a 23 item scale that provide a total score from 0-78 with a lower score indicating greater severity.
Measuring the effects of Nilotinib on Behavior using the Neuropsychiatric Inventory (NPI) | 6 Months
  The NPI is a multi-item instrument to assess psychopathology in Azheimer's disease based on interview with the study partner. The NPI evaluates both the frequency and severity of 10 neuropsychiatric disturbances. Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously) as well as severity (1=mild, 2=moderate, 3=severe). The overall score and the score for each subscale are the product of severity and frequency.
Measuring the effects of Nilotinib on Behavior using the Clinical Assessment of Fluctuation (CAF) | 6 Months
  The CAF consists of seven items of confusional behavior (falls, fluctuation, drowsiness, attention, disorganized thinking, altered level of consciousness, communication), scores for which are summed to provide a severity score for fluctuating confusion ranging from 0 to 21
Measuring the effects of Nilotinib on Behavior using the Irritability-Apathy Scale (IAS) | 6 Months
  The IAS measures apathy and irritability in patients with dementia. The IAS is a 28-item self-administered questionnaire collecting information about different aspects of irritability and apathy utilizing a 0-3 scale for each item to indicate severity. Both a patient and a study partner version can be administered. The IAS will be completed separately by Subjects and Study Partners. A higher total score indicates higher severity , a lower one indicated lower severity.
Measuring the effects of Nilotinib on Behavior using the Problem Behaviors Assessment short form (PBA-s) | 6 Months
  PBA-s is a structured interview in which a trained interviewer rates the frequency and severity of neuropsychiatric symptoms through observation and the reporting of the Subject and Study Partner. Symptoms rated include depressed mood, suicidal ideation, anxiety, irritability, angry or aggressive behavior, apathy, perseverative thinking or behavior, obsessive-compulsive behaviors, delusional or paranoid thinking, hallucinations, and disoriented behavior. Each behavioral problem is rated for both severity and frequency on a 0-4- point scale; severity and frequency ratings are then multiplied to provide an overall score for each symptom.
Measuring the effects of Nilotinib on Motor Function by using the Unified Parkinson's Disease Rating Scale (UPDRS)-I-III. | 6 Months
  UPDRS-I-III is used to follow the longitudinal course of Parkinson's disease. The UPDRS is made up of these sections: Part I: evaluation of mentation, behavior, and mood. Part II: self-evaluation of the activities of daily life (ADLs) Part III: clinician-scored monitored motor evaluation. Part IV: complications of therapy. Part V: Hoehn and Yahr staging of severity of Parkinson's disease. Part VI: Schwab and England ADL scale. The greater the score the higher the severity, the lower the score the lower the severity. The maximum possible UPDRS score is 199.
Measuring the effects of Nilotinib on Motor Function by using the Timed-Up-And-Go (TUG). | 6 Months
  Timed Up and Go (TUG) is an assessment of mobility, balance, walking ability, and fall risk. It measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. This assessment is measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L Pagan, MD, Principal Investigator — Georgetown University
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hebron ML, Lonskaya I, Moussa CE. Nilotinib reverses loss of dopamine neurons and improves motor behavior via autophagic degradation of alpha-synuclein in Parkinson's disease models. Hum Mol Genet. 2013 Aug 15;22(16):3315-28. doi: 10.1093/hmg/ddt192. Epub 2013 May 10. PMID 23666528
- See also: https://sites.google.com/a/georgetown.edu/moussa-lab/lab-members — https://neurology.georgetown.edu/translational_neurotherapeutics